CLINICAL TRIAL: NCT05695742
Title: Smoking Cessation Outcomes and Effective Factors: Maximal Voluntary Breath-holding Time and Exercise Capacity
Brief Title: Smoking Cessation Outcomes and Effective Factors
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Smoking
Record Dates: First submitted 2022-12-26; First posted 2023-01-25 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-01

CONDITIONS: Smoking Cessation
Keywords: smoking; active smoking; pasive smoking; exercise capacity; maximal voluntary breath holding; Fagerstrom
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active smokers: Having smoked at least 1 cigarette per day for at least 2 years.
  Interventions: Other: Active Smoking
- Pasive smokers: Being exposed to secondhand smoke for more than 15 minutes at home, school, office or anywhere in the past year, once a week.
  Interventions: Other: Passive smoker
- Non-smokers: Not being an active or passive smoker.
  Interventions: Other: Non-smoker

INTERVENTIONS:
Other: Active Smoking — Being active smoker
  Groups: Active smokers
Other: Passive smoker — Being exposed to secondhand smoke
  Groups: Pasive smokers
Other: Non-smoker — Not being an active or passive smoker.
  Groups: Non-smokers

SUMMARY:
The study is a cross-sectional-descriptive study. Cases who met the inclusion criteria, agreed to participate in the study voluntarily, were active smokers, passive smokers and non-smokers will be included. The subjects will be given the maximal voluntary breath-hold test, the 6-minute walk test, and the 30-second sit-and-stand test, and will be asked to answer questions about smoking. The physical conditions of the groups will be compared.

DETAILED DESCRIPTION:
The study is a cross-sectional-descriptive study. Cases who met the inclusion criteria, agreed to participate in the study voluntarily, were active smokers, passive smokers and non-smokers will be included. Active smoking, passive smoking status and non-smoker status of the cases will be determined within the framework of the definitions given below.

* Active smoker: Having smoked at least 1 cigarette per day for at least 2 years.
* Passive smoker: Being exposed to secondhand smoke for more than 15 minutes at home, school, office or anywhere in the past year, once a week.
* Non-smoker: Not being an active or passive smoker.

The subjects will be given the maximal voluntary breath-hold test, the 6-minute walk test, and the 30-second sit-and-stand test, and will be asked to answer questions about smoking.The physical conditions of the groups will be compared.

ELIGIBILITY:
Inclusion Criteria for Active Smokers

* Being between the ages of 18-75
* Smoking at least 1 cigarette a day for at least 2 years

Inclusion Criteria for the Passive Smoker Group

* Being between the ages of 18-75
* Being exposed to cigarette smoke for more than 15 minutes at home, school, office or anywhere in the last year, once a week.

Inclusion Criteria for the Non-Smoker Group

* Being between the ages of 18-75
* Not being an active or passive smoker

Exclusion Criteria:

* Having any disease that prevents him from doing exercise tests
* Not signing the voluntary informed consent form

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Active, pasive smoker and non-smoker volunters
Sampling Method: Probability Sample
Enrollment: 893 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Six-minute walking test | 1 day
  The subject will be asked to walk for 6 minutes on a flat surface of 30 meters and the distance covered will be recorded. The test will be performed in accordance with the American Thoracic Society guidelines
Maximal voluntary breath-hold time | 1 day
  The maximum voluntary breath-hold test is a quick and simple test that consists of measuring the apnea time after a deep inspiration. The clinical utility of this test has been proven in certain respiratory pathologies. In the test, the subject will be seated in a chair with back support, a deep inspiration will be asked, and the breath-holding time will be recorded in seconds. The test will be repeated three times with sufficient rest periods in between, and the longest time will be analyzed.

SECONDARY OUTCOMES:
Thirty Seconds Sit and Stand test | 1 day
  During the test, the individual performs the sit-stand-sit maneuver from a standard height chair within 30 seconds without using his arms as much as possible. The number of sitting and standing up during this period is recorded.
Fagerstrom Nicotine Addiction Test | 1 day
  Dependence analysis will be performed on smokers according to the Fagerström nicotine addiction test and the scales for evaluating the psychological dependence of cigarettes. It is a six-question questionnaire created by revising the Fagerstrom tolerance questionnaire. In the scoring made according to the answers given to the questions, 0-2 points is called very mild addiction and 8-10 points is called very severe addiction
Evaluation scale of psychological dependence on cigarette | 1 day
  It is a scale used in the evaluation of psychological dependence on cigarettes. The possible scores range from 25 to 75. As the scale score increases, the degree of psychological dependence increases; Scoring; 25-41 score: mildly addicted 42-58 score: moderate addiction

CONTACTS AND LOCATIONS:
Overall Officials: ESRA PEHLİVAN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)